CLINICAL TRIAL: NCT05455450
Title: Randomised Feasibility Study of Eye Movement Desensitisation and Reprocessing Therapy (EMDR) for Functional Neurological Disorder (FND)
Brief Title: Eye MOvement DesensItisation and Reprocessing Therapy (EMDR) for FunctIonal Neurological Disorder (FND)
Acronym: MODIFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South West London and St George's Mental Health NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: COPS1001
Record Dates: First submitted 2022-06-14; First posted 2022-07-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Functional Neurological Symptom Disorder
Keywords: Functional neurological disorder, FND
MeSH Terms: conditions — Conversion Disorder; Frontonasal dysplasia | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into EMDR (plus neuropsychiatric care; NPC) or NPC. A stratified block randomisation will be used to ensure similar numbers of patients with predominant functional seizures or functional motor disorder, and PTSD/non-PTSD are relatively equal across arms.
Who Masked: Outcomes Assessor
Masking Description: The assessing RA and project statistician will be blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR + NPC (Experimental): 8-16 eye movement desensitisation and reprocessing therapy (EMDR) sessions, plus 1 month follow up session after the therapy has ended. Participants will also attend neuropsychiatric follow-up appointments as part of standard medical care.
  Interventions: Other: Eye movement desensitisation and reprocessing therapy; Other: Neuropsychiatric care
- Neuropsychiatric Care (NPC) (Other): Standard medical care
  Interventions: Other: Neuropsychiatric care

INTERVENTIONS:
Other: Eye movement desensitisation and reprocessing therapy — Up to 16 EMDR sessions (minimum of 8 sessions), and 1-month follow-up session, as well as attending neuropsychiatric appointments (NPC). Participants will be given the choice of attending EMDR physically face-to-face or virtually via a video-consultation platform. Sessions will normally be attended weekly, with treatment completed within 6 months. Sessions will be 60-90 minutes long. EMDR will follow the standard 8-phase protocol, with additions so that it is tailored for FND presentations. The FND-specific EMDR therapy protocol has been developed for the trial by the chief investigator.
  Other Names: EMDR
  Arms: EMDR + NPC
Other: Neuropsychiatric care — Standard medical care consisting of 1-3 30 minute appointments with neuropsychiatrist over the course of the 9-month trial period.

SUMMARY:
Functional Neurological Disorder (FND) is a problem with the functioning of the nervous system and how the brain and body send and receive signals, rather than due to neurological disease or injury. This causes a range of neurological symptoms such as seizures, shaking, weakness, and paralysis. The symptoms are associated with significant distress and disability. Treatment for FND in the United Kingdom is limited, and the evidence-base for treatment is poor, despite it being a common presentation. A psychological therapy called cognitive-behavioural therapy has been found to be beneficial, but it does not help everyone. EMDR is an effective treatment for posttraumatic stress disorder, but it can also be helpful with other conditions. There is a small amount of case study evidence that EMDR can be useful at treating FND, but proper scientific evaluation is needed.

This research aims to evaluate the possibility of delivering, and potential benefit, of EMDR for FND. If the study shows that it is feasible and potentially beneficial, a larger trial will be designed. The study will recruit 50 participants who have specific functional neurological symptoms: weakness, walking difficulties, jerks, shaking, and/or seizures from a Neuropsychiatry Service. Participants will be allocated to EMDR, and routine medical appointments, or routine medical appointments alone. Allocation will be carried out by a computer programme. Those allocated to EMDR will be offered 8-16 weekly therapy sessions, completed within 6 months, and follow-up session 1 month after therapy has ended. Participants will be able to choose whether to attend therapy in-person or via an online video conferencing platform. Participants will complete questionnaires regarding health-related functioning, FND, mental health, and healthcare utilisation. These questionnaires will be completed at the beginning, 3 months, 6 months, and 9 months.

Some participants will attend interviews about experiences of treatment.

DETAILED DESCRIPTION:
Background:

Functional neurological disorder (FND) refers to an involuntary loss of control over and/or aberrant perception of the body. Common presenting symptoms are functional (non-epileptic) seizures, and functional motor disorder, e.g. walking difficulties, weakness, or tremor. Treatment in the United Kingdom is inconsistently available, and there is inequity of care compared to other neurological conditions. There are no established standards of care for this patient group. FND is associated with large health- and social-care costs. Greater access to effective treatments would lead to reduced distress and disability for patients with FND; and reduce unnecessary costs to the NHS.

This research proposes using eye-movement desensitisation and reprocessing therapy (EMDR) as a treatment for FND. EMDR is an evidence-based treatment for post-traumatic stress disorder (PTSD), but its use for other conditions is growing. A FND-specific EMDR protocol will be developed and tested, and if the intervention proves feasible with promising clinical outcomes, progression to a substantive study could take place.

Aims and Objectives:

I. Test the acceptability and feasibility of an FND-specific EMDR intervention protocol, delivered physically or virtually.

II. Investigate the value of a range of outcome measures, to determine the outcome measure with greatest symptom improvement and the required sample size, for a substantive RCT.

III. Carry out semi-structured interviews with participants and therapists to explore experiences of EMDR and the trial; informing the intervention and design for a substantive trial.

Methods:

50 adult patients with a diagnosis of FND will be recruited via a Neuropsychiatry Service. The study will be a single-blind randomised controlled trial (RCT) with two arms: EMDR (plus standard neuropsychiatric care; NPC) and standard NPC. The two groups will be compared at baseline (T0), 3 months (T1), 6 months (T2), and 9 months (T3). Measures of feasibility include safety, recruitment, retention, and treatment adherence and acceptability. Clinical outcome measures assess health-related functioning/quality of life, FND, depression, anxiety, PTSD, dissociation, service-utilisation and other costs. Patient-rated improvement and satisfaction will also be assessed. Feasibility outcomes will be summarised using descriptive statistics. Exploratory analyses using (linear/logistic) Mixed Effect Models will examine the rate of change in intervention and control groups' clinical outcome measures across the four time-points.

After the intervention period, a sample of participants, and clinicians, will be invited to attend semi-structured interviews on trial experiences. The interviews will be analysed using reflexive thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Predominant diagnosis of functional seizures and/or functional motor disorder, with diagnosis confirmed by neurologist
2. Aged 18 years or over
3. Capacity to consent
4. Willingness to attend regular psychological therapy sessions
5. Reporting at least 1 traumatic event on the International Trauma Exposure Measure

Exclusion Criteria:

1. Non-English speaking
2. Current ongoing adversity that is likely to interfere with psychological therapy, e.g. domestic violence, homelessness, unresolved compensation claim/litigation
3. Predominant diagnosis of Borderline Personality Disorder*
4. Predominant diagnosis of chronic pain condition*, e.g. fibromyalgia
5. Predominant diagnosis of chronic fatigue syndrome*
6. Diagnosis of a psychotic disorder
7. Diagnosis of Dissociative Identity Disorder or score in clinical range on "identity disturbance" subscale of Multiscale Dissociation inventory
8. Uncontrolled epileptic seizures
9. Diagnosis of an eating disorder
10. Current severe self harm or strong suicidal ideation that requires secondary care mental health services input
11. Current alcohol or drug harmful-use or dependence
12. Current diazepam use exceeding the equivalent of 10mg per day
13. Currently attending individual psychological therapy focused on functional neurological disorder or other specialist functional neurological disorder-specific treatment such as inpatient/outpatient multi-disciplinary treatment or intensive functional neurological disorder-specific physiotherapy

    * Comorbid diagnosis is acceptable, as long as functional neurological disorder is the predominant difficulty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 months (recruitment stage)
  Percentage of potentially eligible participants attending screening interview
Intervention adherence | 18 months (intervention stage)
  Percentage of participants randomised to EMDR+NPC who complete therapy
Outcome measures completion | 12 months (9-month follow-up stage)
  Percentage of participants who complete outcome measures at all 4 time points

SECONDARY OUTCOMES:
EQ-5D-5L | 4 time points over 9 months (trial period)
  Brief health questionnaire
Ecological Momentary Assessment (EMA) of FND symptoms | 4 time points over 9 months (trial period)
  Using an App, FND symptoms will be rated in terms of frequency, severity, interference with daily functioning, associated distress and preoccupation with
PHQ-9 | 4 time points over 9 months (trial period)
  Self-rated measure of depression
GAD-7 | 4 time points over 9 months (trial period)
  Self-rated measure of anxiety
International Trauma Questionnaire (ITQ) | 4 time points over 9 months (trial period)
  Measure of PTSD and Complex PTSD
Multiscale Dissociation Inventory | 4 time points over 9 months (trial period)
  Measure of dissociation
Adult Service Use Schedule (AD-SUS) | 2 time points over 9 months (trial period)
  Self-report measure of service use
World Health Organisation Disability Assessment Schedule (WHODAS 2.0) | 4 time points over 9 months (trial period)
  Health-Related Quality of life/functioning measure

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R Cope, DClinPsy, Principal Investigator — South West London & St. George's Mental Health NHS Trust
Locations (2):
- United Kingdom (2):
  - South West London & St George's NHS Trust, London
  - Neuropsychiatry Service, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cope SR, Smith JG, El-Leithy S, Vanzan S, Hogwood P, Golder D, Turner KJ, Crowley M, Billings J, Pick S, Pentland C, Edwards MJ. Randomised feasibility study evaluating eye movement desensitisation and reprocessing therapy for functional neurological disorder (MODIFI). J Neurol. 2025 Jul 8;272(8):493. doi: 10.1007/s00415-025-13219-5. PMID 40627223
- [Derived] Cope SR, Smith JG, El-Leithy S, Vanzan S, Pentland C, Pick S, Golder D, Hogwood P, Turner K, Billings J, Edwards MJ. MODIFI: protocol for randomised feasibility study of eye-movement desensitisation and reprocessing therapy (EMDR) for functional neurological disorder (FND). BMJ Open. 2023 Jun 2;13(6):e073727. doi: 10.1136/bmjopen-2023-073727. PMID 37270188